CLINICAL TRIAL: NCT06893003
Title: A Pilot Study on Cost and Other Implementation Factors Comparing Telehealth and In-Person Therapy Service Delivery Following NICU Discharge
Brief Title: A Pilot Study Comparing Telehealth and In-Person Therapy Service Delivery Following NICU Discharge
Acronym: BabyBridge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Roberta Pineda, Associate Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AOTFIR21; AOTFIR21 (Other Grant/Funding Number: American Occupational Therapy Foundation)
Record Dates: First submitted 2025-03-07; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Prematurity Complications; NICU Infants; Early Intervention; Telehealth
Keywords: Baby Bridge; Early intervention; Telehealth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telehealth Baby Bridge model (Experimental): For those assigned to the telehealth Baby Bridge group, a first telehealth visit will be scheduled within one week of discharge, and weekly telehealth visits will be scheduled thereafter. However, parents will be informed that in-person visits are an option when needs arise. Adaptations from a telehealth visit to an in-person visit will be made in the event of therapist clinical judgment due to the medical complexity or feeding/tonal abnormalities of the infant and parent preference or rapport building. Visit adaptations will be tracked along with the reasoning for them.
  Interventions: Other: Baby Bridge
- In-Person Baby Bridge model (Active Comparator): For those assigned to the in-person Baby Bridge group, the first visit will be scheduled in the home within one week of NICU discharge, and attempts will be made to see the infant weekly in the home environment for a one-hour therapy session. Scheduled visits will be confirmed with families via text messaging the day before each visit. Visits will be rescheduled to telehealth in the event of therapist illness, parent preference or parent/child illness, or distance or therapist schedule limitations. Changes of visits from in-person to telehealth will be tracked along with their reasoning.
  Interventions: Other: Baby Bridge

INTERVENTIONS:
Other: Baby Bridge — The Baby Bridge program is an evidence-based implementation strategy aimed at enhancing early and continuous therapy services following NICU discharge for infants with alterations in neurodevelopment. The Baby Bridge program utilizes an occupational or physical therapist to see the infant and family in the NICU prior to discharge, complete a comprehensive neurodevelopmental and feeding assessment to inform targeted interventions, and provide early therapy services in the home environment within one week of discharge and weekly thereafter, until other community-based services commence. While most of the program occurs after NICU discharge, a hallmark of the Baby Bridge program is that families establish rapport with the therapist while the infant is still in the NICU. The therapist also educates the family on ways to support their infant's development between sessions and offers support and assistance during the transition from hospital to home.

SUMMARY:
20 high-risk parent-infant dyads hospitalized in a 58-bed level IV NICU will be randomized to either receive Telehealth or in-person Baby Bridge services. Baby Bridge is a program to bridge the gap between NICU discharge and initiation of community-based early intervention services. Weekly therapy services are provided in the child's home, either via telehealth or in-person. An in-person evaluation in the NICU is attempted for each child prior to NICU discharge. Cost, adoptability, feasibility, adaptations, and acceptability amongst caregivers will be compared between the two groups.

DETAILED DESCRIPTION:
Participants and setting

Participants include 20 high-risk parent-infant dyads hospitalized at CHLA. Enrolled infants and families will be randomized to receive Baby Bridge services either through telehealth or in-person visits. Parent-infant dyads will be enrolled at least 2 days before NICU discharge to enable rapport to be established (between the Baby Bridge therapist and family) through a visit to the NICU when possible and via telephone, text or email messaging when an in-person visit is not possible prior to discharge. This first contact will be attempted to be in-person in the NICU for both the telehealth and in-person groups. Enrolled infants and families will then have a Baby Bridge telehealth or in-person visit scheduled within one week of discharge (depending on their group assignment). Subsequent individual weekly visits will be adapted to in-person or telehealth (varying from assigned group) when needed or deemed appropriate (requested by the family or therapist or when an in-person visit is felt to improve the quality of the therapy session). Weekly Baby Bridge programming will be conducted until other therapy through the state-wide early intervention program commences, as in the infant begins receiving therapy services as recommended. Investigators will also track rates of enrollment, rates and reasons for any cancellations, and completion of the program (defined as being seen until community-based early intervention services commenced). Infants will be withdrawn if they are transferred to another hospital prior to discharge or if they are readmitted to the hospital and additional contact was not possible or feasible.

Sociodemographic and medical data will be collected from the electronic medical record for each dyad enrolled to better understand differences between groups as well as to define sample characteristics. Sociodemographic factors collected will include: infant race, insurance type (public or private), maternal age, number of siblings, home distance from the hospital, and categorization of home residence (urban with <3,000 people per square mile, suburban with between 1,000 and 3,000 people per square mile, or rural with <1,000 people per square mile). Medical factors collected will include: estimated gestational age at birth, the primary condition of the infant (congenital anomaly, preterm birth, or neurological condition not related to preterm birth or congenital anomaly), number of days of endotracheal intubation, number of days of hospitalization, and whether or not the infant was orally feeding at time of hospital discharge.

In-person group assignment For those assigned to the in-person Baby Bridge group, the first visit will be scheduled in the home within one week of NICU discharge, and attempts will be made to see the infant weekly in the home environment for a one-hour therapy session. Scheduled visits will be confirmed with families via text messaging the day before each visit. Visits will be rescheduled to telehealth in the event of therapist illness, parent preference or parent/child illness, or distance or therapist schedule limitations. Changes of visits from in-person to telehealth will be tracked along with their reasoning.

Telehealth group assignment For those assigned to the telehealth Baby Bridge group, a first telehealth visit will be scheduled within one week of discharge, and weekly telehealth visits will be scheduled thereafter. However, parents will be informed that in-person visits are an option when needs arise. Adaptations from a telehealth visit to an in-person visit will be made in the event of therapist clinical judgment due to the medical complexity or feeding/tonal abnormalities of the infant and parent preference or rapport building. Visit adaptations will be tracked along with the reasoning for them.

Implementation outcomes The primary outcome of interest for this study will be cost difference between telehealth and in-person visits of the Baby Bridge program. Investigators also plan to investigate implementation outcomes of adoptability (enrollment rate), feasibility (whether program tenets were followed), adaptations, and acceptability (parent satisfaction).

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized in the NICU for >7 days
* Received a referral for early intervention at time of NICU discharge
* Was referred to program at least 48 hours before NICU discharge

Exclusion Criteria:

* Chronological age >6 months at time of NICU discharge
* Non-English speakers
* Those discharging home to a different state/country

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2025-03-03 (Actual)

PRIMARY OUTCOMES:
Cost of the Baby Bridge program | From first Baby Bridge visit to last Baby Bridge visit for each infant (approx 12 weeks but varies significantly between infants)
  For the purposes of this project, we estimated costs associated with each Baby Bridge visit. We did not assess cost across group assignment, due to the allowed adaptations to each visit type. Cost was defined in relation to the organizational cost of providing Baby Bridge visits and included the time that the therapist spent conducting therapy sessions (billable time), administrative time (documentation, communication with families), driving (for in-person visits), and mileage reimbursement.

SECONDARY OUTCOMES:
Adoptability of the Baby Bridge program | From first Baby Bridge visit to last Baby Bridge visit for each infant (approx 12 weeks but varies significantly between infants
  Number of infants referred, approached, and enrolled. Adoption was operationalized to include the total number of infants approached versus enrolled (enrollment rate).
Feasibility of the Baby Bridge program - Timing | From first Baby Bridge visit to last Baby Bridge visit for each infant (approx 12 weeks but varies significantly between infants
  We captured timing (if the first visit was conducted within one week of discharge); average time from NICU discharge to first Baby Bridge visit); frequency of visits; rate and reasons for any therapy visit cancellations; the completion rates (percentage of enrolled infants who completed programming); and the timing of transition to community-based therapy. Feasibility was defined a priori as all Baby Bridge visits attempted within the first week, infants seen at least 3 visits per month while in the program, and that 80% would be successfully transitioned to early intervention programming.
Feasibility of the Baby Bridge program - Frequency | From first Baby Bridge visit to last Baby Bridge visit for each infant (approx 12 weeks but varies significantly between infants
  Frequency of Baby Bridge visits, as well as rate and reasons for any therapy visit cancellations; the completion rates (percentage of enrolled infants who completed programming); and the timing of transition to community-based therapy. Feasibility was defined a priori as all Baby Bridge visits attempted within the first week, infants seen at least 3 visits per month while in the program, and that 80% would be successfully transitioned to early intervention programming.
Feasibility of the Baby Bridge program - Completion rate | From first Baby Bridge visit to last Baby Bridge visit for each infant (approx 12 weeks but varies significantly between infants
  Completion rates (percentage of enrolled infants who completed programming); and the timing of transition to community-based therapy. Feasibility was defined a priori as all Baby Bridge visits attempted within the first week, infants seen at least 3 visits per month while in the program, and that 80% would be successfully transitioned to early intervention programming.
Feasibility of the Baby Bridge program - Timing of transition | From first Baby Bridge visit to last Baby Bridge visit for each infant (approx 12 weeks but varies significantly between infants
  Timing of transition to community-based therapy
Adaptations to the Baby Bridge program | From first Baby Bridge visit to last Baby Bridge visit for each infant (approx 12 weeks but varies significantly between infants
  Proportion of visits conducted via telehealth in the telehealth group and proportion of visits that occurred in-person in the in-person group. Reasoning for such adaptations was tracked as described above in the telehealth and in-person assignment sections.
Acceptability of the Baby Bridge program | From first Baby Bridge visit to last Baby Bridge visit for each infant (approx 12 weeks but varies significantly between infants
  Upon completion of the Baby Bridge program, parents were asked to complete the Baby Bridge Parent Survey to query their perceptions about Baby Bridge programming. Survey questions were loaded into REDCap and administered electronically through a shared link to a REDCap survey. Parent satisfaction was measured based on a sum (possible range of 0-10) of the questions on the survey.

CONTACTS AND LOCATIONS:
Overall Officials: Roberta Pineda, PhD, OTR/L, Principal Investigator — University of Southern California
Locations (2):
- United States (2):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - University of Southern California, Los Angeles, California

IPD SHARING:
Plan to Share IPD: No
Pilot study; small enough sample that even diagnoses could be considered PHI

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-03-07): https://cdn.clinicaltrials.gov/large-docs/03/NCT06893003/Prot_SAP_000.pdf